CLINICAL TRIAL: NCT04515069
Title: Survival of a Recent Polymer- Infiltrated Ceramic Network Laminate Veneer Material Using Aesthetic Preevaluative Temporary (APT) Technique Versus Traditional Technique in the Aesthetic Zone:Randomized Clinical Trial
Brief Title: Survival of Hybrid Laminate Veneers Using Two Different Tooth Preparation Techniques:Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Attia, Assistant Lecturer, Fixed Prosthodontics Department, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 151021
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Discoloration, Tooth; Malformed Tooth; Diastema
Keywords: veneers; hybrid ceramics; CAD/CAM; tooth preparation techniques; USPHS criteria
MeSH Terms: conditions — Tooth Discoloration; Tooth Abnormalities; Diastema | interventions — Sensitivity Training Groups; Tooth Preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization was done using a computer generated 2 column list by the aid of Random.org in a 1:1 ratio. Allocation concealment was achieved using numbered cards in opaque sealed envelopes. Aluminium foil was placed inside the envelope to render the envelope impermeable to intense light. These envelopes were placed in a box and each participant was allowed to grasp one envelop the day of operation. Allocation concealment was performed by an investigator with no clinical involvement in the trial. This study is a single blinded study as the assessor was blinded to the assigned study groups. Blinding of the participants was not applicable as one of the techniques required extra visits. Blinding of the operator was not applicable as one clinician performed the tooth preparation in both techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional technique for tooth preparation. (Active Comparator): Tooth preparation performed directly on the tooth structure
  Interventions: Procedure: traditional technique of tooth preparation
- Aesthetic preevaluative temporary technique (Active Comparator): Aesthetic pre-evaluative temporary (APT) was fabricated according the planned wax-up. Once the APT was approved both aesthetically and functionally, tooth preparation was performed through the APT.
  Interventions: Procedure: aesthetic preevaluative temporary technique for tooth preparation

INTERVENTIONS:
Procedure: traditional technique of tooth preparation — Depth cutter wheels of predetermined depths (Komet, Germany) were used to perform the preparation directly on the tooth structure.
  Depth cuts were performed on the labial surface using depth cutter wheels (Komet, Germany) with radius of 0.3 mm and 0.5 mm which is directly related to the thickness of the laminate veneers in the cervical and incisal one thirds respectively. Then islands of tooth structure between depth orientation grooves were removed.
  Proximal reduction:
  The interproximal reduction was completed just labial to the contact areas using a round end tapered diamond stone (Mani, Japan), and polishing was performed using polishing strips (Sof-Lex, 3M ESPE, Seefeld, Germany).
  Incisal reduction:
  Vertical depth grooves were created. Then, the round end tapered diamond stone (Mani, Japan)was used to create 1.5 mm incisal butt joint preparation.
  Then, finishing and polishing of tooth preparation was performed.
  Other Names: Group T
  Arms: Traditional technique for tooth preparation.
Procedure: aesthetic preevaluative temporary technique for tooth preparation — The data obtained from digital smile design was used for construction of the diagnostic wax-up. The wax-up was then be transferred to the mouth using a silicone index, creating the aesthetic pre-evaluative temporary (APT). The APT was tested esthetically and functionally. Once approved by the operator and the patient, tooth preparation was performed through the APT. Depth cuts were performed similar to those performed in the traditional preparation with the difference of being prepared on the aesthetic pre-evaluative temporary instead of directly on the dental structure. Using tapered stone with round end (Mani, Japan), islands of tooth structure between depth orientation grooves were removed.
  Proximal reduction, Incisal reduction Finishing and polishing of tooth preparation were carried out using the same technique as in the Group T with the difference of being performed through the APT, resulting in minimal tooth preparation
  Other Names: Group A
  Arms: Aesthetic preevaluative temporary technique

SUMMARY:
The aim of this study was to evaluate the survival of laminate veneers constructed using a recent polymer-infiltrated ceramic network material following the aesthetic pre-evaluative temporary (APT) technique of tooth preparation in comparison to traditional technique.

DETAILED DESCRIPTION:
Six recruited patients (4 females, 2 males; ranging from: 20-30 years old and with mean age 24.6 years), who needed indirect laminate veneer restorations were included in this study. Patients were selected from the outpatient clinic of the Department of Fixed Prosthodontics,Faculty of Dentistry, Cairo University The participants received a total of 54 laminate veneers between April 2017 and February 2018. Written informed consent was acquired from all participating patients. Randomization was done using a computer generated 2 column list by the aid of Random.org in a 1:1 ratio. Allocation concealment was achieved using numbered cards in opaque sealed envelopes. Aluminium foil was placed inside the envelope to render the envelope impermeable to intense light. These envelopes were placed in a box and each participant was allowed to grasp one envelop the day of operation. Allocation concealment was performed by an investigator with no clinical involvement in the trial. This study is a single blinded study as the assessor was blinded to the assigned study groups. Blinding of the participants was not applicable as one of the techniques required extra visits. Blinding of the operator was not applicable as one clinician performed the tooth preparation in both techniques.A total of 54 laminate veneers were divided into two equal groups (n=27) according to the technique of tooth preparation: group T: traditional technique and group A: aesthetic pre-evaluative temporary technique. VITA ENAMIC material was used for CAD/CAM construction of laminate veneers. Cementation was performed using a light cured resin cement. The laminate veneers were evaluated at baseline, after 3, 6 and 12 months according to the modified United States Public Health Service (USPHS) criteriea. The data was collected, tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Patients consulting the outpatient clinic of the department of Fixed Prosthodontics, Faculty of Dentistry, Cairo University.
  * Able to tolerate necessary restorative procedures.
  * Provide written consent.
  * Accepts the one year follow-up period.

Tooth related criteria:

* Malaligned and malformed teeth in the aesthetics zone
* Multiple spacing
* Diastema
* Slightly and moderately discolored teeth
* Good oral hygiene

Exclusion Criteria:

Patient-related criteria:

* Medically compromised patients, as they would not be able to attend multiple appointments or might require special management.
* Uncooperative patients, who would not abide by the instructions or attend the appointments.

Tooth related criteria:

* Deciduous teeth; as the study was targeting only permanent teeth.
* Teeth with previous restorations, which might add another variable to the study (type of old restorative material, extent of recurrent caries). This could also affect the bond of laminate veneers to tooth structure.
* Patients with parafunctional habits, large restorations, or excessive tooth wear.
* Initially, scaling and polishing was performed. Patients were instructed on improving their oral hygiene and maintaining effective plaque control. However, if their gingival health did not improve, they were excluded from the study.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Survival of laminate veneers using modified USPHS | 1 year
  Patients were called back after 1 week as the baseline to assess the veneer restorations. Assessment was carried out by an experienced observer blinded to the assigned study group for each patient. Laminate veneers were examined at baseline, after 3, 6 and 12 months according to the modified United States Public Health Service (USPHS) criteriae and the USPHS scores of Alfa, Bravo and Charlie were used for rating . Patients were also questioned about possible post-operative complaints. Digital photographs were made after placement of the veneers and during follow-up sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa Zaghloul, PhD, Study Director — Professor of Fixed Prosthodontics, Misr International University
Locations (1):
- Yara Attia, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Clinical Study Report
Supporting Information: CSR
Time Frame: starting 6 months after publication
Access Criteria: Data will be available for students and researchers